CLINICAL TRIAL: NCT04307368
Title: The Impact of Dietary Treatment Using a Low FODMAP Diet on the Occurrence of Selected Intestinal Bacteria and the Clinical Condition of Patients With Irritable Bowel Syndrome
Brief Title: The Impact of Dietary Treatment in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Diana Wasiluk, Principal Investigator, Medical University of Bialystok
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-I-002/389/2015
Record Dates: First submitted 2020-02-25; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; diet
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FODMAP diet (Experimental): Patients with IBS. Interventions: 8 weeks of diet low in fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP)
  Interventions: Other: FODMAP diet
- Elimination-rotational diet (Experimental): Patients with IBS. Interventions: During the patient's first visit an IgG antibody titration test against specific nutrients will be performed to determine food hypersensitivity. Based on the results of the obtained food panels, patients will be offered an elimination-rotational diet for a period of 8 weeks.
  Interventions: Other: Elimination-rotational diet
- Classic diet (Experimental): Patients with IBS. Interventions: 8 weeks of classic diet treatment (recommended by the gastroenterologist who supervises them).
  Interventions: Other: Classic diet

INTERVENTIONS:
Other: FODMAP diet — 8 weeks of diet low in fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP)
  Arms: FODMAP diet
Other: Elimination-rotational diet — During the patient's first visit an IgG antibody titration test against specific nutrients will be performed to determine food hypersensitivity. Based on the results of the obtained food panels, patients will be offered an elimination-rotational diet for a period of 8 weeks.
  Arms: Elimination-rotational diet
Other: Classic diet — 8 weeks of classic diet treatment (recommended by the gastroenterologist who supervises them).
  Arms: Classic diet

SUMMARY:
The obtained results are likely to determine whether changes in the diet of patients with irritable bowel syndrome will affect their nutritional status. They will also allow you to assess whether dietary treatment will affect the resolution or alleviation, or severity of disease symptoms in IBS. The test results can be used in clinical practice.

Participation in the study does not carry any risk of complications associated with undergoing a medical experiment.

DETAILED DESCRIPTION:
This is a randomized, parallel study that includes 1 initial visit and 1 final visit, separated by 8 weeks of diet. The investigators enrolled 73 women in the study, who met the criteria for inclusion in the study, to determine whether changes in the diet of patients with irritable bowel syndrome will affect their nutritional status. At the initial and final visit (after 8 weeks) in all patients, anthropometric measurements, body composition, an interview questionnaire concerning the symptoms of the disease was performed, the intensity of abdominal pain was assessed, the life quality of patients on the IBS-QOL scale was assessed, the calprotectin concentration in the stool was determined and the questionnaire regarding the quantitative assessment of diet was performed. The study population was divided using simple lottery into 3 groups with different dietary treatment for 8 weeks: group 1 - 26 patients - diet with low content of easily fermenting carbohydrates (FODMAP), group 2 - 21 patients - an elimination-rotation diet, and group 3 - (control) - 26 patients - classic diet treatment (recommended by the leading gastroenterologist).

ELIGIBILITY:
Inclusion Criteria:

1. patients with irritable bowel syndrome (mixed) according to Rome III Criteria, in whom the gastroenterologist does not find any other gastrointestinal diseases that may affect this study
2. patients who understand the purpose and nature of the study, agree to its terms and give informed written consent before entering the study
3. who are physically and mentally able to participate in the study and express their will to cooperate

Exclusion Criteria:

1. patients who use strong opioid and psychotropic drugs: barbiturates
2. patients who take part in another clinical trial related to the treatment of gastrointestinal diseases or dietary therapy within 90 days prior to inclusion in this study
3. patients who have a pacemaker or heart defibrillator implanted and metal endoprostheses (due to the used body composition test method (BIA - Bioelectrical Impedance Analysis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Comparative analysis of selected clinical symptoms of IBS patients before and after 8 weeks of nutritional intervention. | 8 weeks
  During the first visit, each applicant will receive a detailed interview on sociodemographic characteristics, lifestyle and professional work. The interview questionnaire contains questions about the most common symptoms of the disease (including abdominal pain, flatulence, stool disorders).
Assessment of intestinal inflammation in patients with irritable bowel syndrome (before and after 8 weeks of using the recommended diet). | 8 weeks
  Intestinal inflammation was assessed by faecal calprotectin. At the first visit, each patient must bring a stool sample to assess calprotectin levels. The test will be carried out normalized and certified by Elisa.
Comparative analysis of the quality of life of IBS patients before and after 8 weeks of nutritional intervention. | 8 weeks
  The current quality of life for patients with irritable bowel syndrome will be assessed using the IBS-QOL (Irritable Bowel Syndrome-Quality Of Life Questionnaire); total score between 34 -170 points, the highest sum means the most reduced quality of life.
Comparative analysis of the nutritional value of diets used before the study and after 8 weeks of dietary treatment using the FODMAP diet, elimination-rotation and conventional. | 8 weeks
  Quantitative diet assessment was based on a 24h diet recall from 3 days preceding the study. The respondents estimated the amount of each food and ingredient consumed. The results from each patient were averaged in accordance with the adopted recommendations of the Institute of Food and Nutrition in Warsaw and the nutritional value of daily food rations was analyzed using Dieta 5.0 software calculating the average intake of the energy, nutrients, vitamins, minerals, cholesterol and dietary fibre.
Individually calculated Body Mass Index | 8 weeks
  Individually calculated BMI (Body Mass Index) - this is the ratio obtained by dividing the body weight in kilograms by the square of the height in meters
Individually calculated Waist-Hip Ratio | 8 weeks
  Individually calculated WHR (Waist-Hip Ratio) - coefficient resulting from dividing the waist circumference by the hip circumference (measurements made in centimeters).
Assessment of nutrients causing food hypersensitivity (IgG1-3) | 8 weeks
  The baseline reaction of alimentary IgG1-3 in blood serum was measured in μg/ml in the ranges: <7.5 μg/ml - not elevated, ≥7.5 μg/ml - increased and ≥20.0 μg/ml - significantly increased.
Assessment of body composition | 8 weeks
  Assessment of body composition of subjects tested using the bioelectroimpedance method (MALTRON BioScan 920-2 by Maltron International LTD).
Pain intesity | 8 weeks
  Pain intensity will be assessed using the VAS (Visual Analogue Scale) numerical scale; total score between 0 -10 points, the higher the value the stronger the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Wasiluk, MS, PhD, Principal Investigator — Medical University of Bialystok

IPD SHARING:
Plan to Share IPD: No